CLINICAL TRIAL: NCT07170293
Title: An Exploratory, Prospective, Single Arm, Open Label, Single Center, Basket, Phase II Clinical Study of Tunlametinib (HL-085) in Patients With NRAS Mutant Non-melanoma Refractory Solid Tumors
Brief Title: Phase II Trial of Tunlametinib in Patients With NRAS Mutant Non-melanoma Refractory Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN-CANCER-NRAS-HL-085
Record Dates: First submitted 2025-09-06; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Solid Cancers
Keywords: NRAS; Tunlametinib; MEK

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tunlametinib (HL-085) (Experimental): Patients with NRAS Mutant Non-melanoma Refractory Solid Tumors.
  Interventions: Drug: Tunlametinib

INTERVENTIONS:
Drug: Tunlametinib — Do not chew, dissolve or open the capsule. If you miss a dose of medication, you can take the missed dose 8 hours before the next dose. If the time until the next medication is less than 8 hours, it is not recommended to take it again. Every 21 days for one cycle, subjects will use the investigational drug until the treatment termination criteria specified in the protocol are met. The recommended dosage for the first dose reduction is 9mg, twice daily. The recommended second dose reduction is 6mg, twice daily.

SUMMARY:
This study is a single cohort, open label exploratory clinical trial aimed at observing and evaluating the efficacy and safety of Tunlametinib (HL-085) in the treatment of refractory solid tumors with advanced metastatic non melanoma. It is expected that the ORR of Tunlametinib (HL-085) treatment can reach 20%. According to the literature results, the experimental group rate is 0.2 and the target value rate is 0.02. If the bilateral alpha is 0.05 and the beta is 0.2, the sample size is calculated as 12 cases in the experimental group. Considering a 20% dropout rate, a total of 15 cases are required.

DETAILED DESCRIPTION:
Members of the RAS gene family, including KRAS, NRAS, and HRAS, can participate in promoting cell metabolism, proliferation, survival, growth, and angiogenesis through the PIK3CA/AKT and RAS/RAF/MAPK signaling pathways downstream of the EGFR tyrosine kinase receptor. Mutations in these genes can lead to sustained activation of downstream signaling pathways, resulting in abnormal cell proliferation and differentiation, which is closely related to the occurrence and development of cancer. The frequency of NRAS gene changes (including CNV and SNV variations) in 10000 patients with advanced metastatic tumors included in the MSK-IMPACT cohort was approximately 3%, with melanoma, thyroid cancer, thymic tumor, primary lesion unknown cancer, and colorectal cancer ranking among the top 5 cancers. At the same time, a large number of domestic studies have shown that the frequency of NRAS gene changes (including CNV and SNV variations) is about 2%, among which the top 5 cancers are melanoma, thyroid cancer, gastrointestinal neuroendocrine tumors, endometrial cancer, and primary lesion unknown cancer. This study is an open exploratory clinical trial aimed at observing and evaluating the efficacy and safety of Tunlametinib in the treatment of non-melanoma refractory solid tumors with NRAS mutations.

ELIGIBILITY:
Exclusion Criteria:

1. Have had other malignant tumors in the past 2 years (excluding tumors with low malignancy such as basal cell carcinoma, squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma, etc. that have undergone radical treatment) or have been diagnosed with melanoma;
2. Moderate or greater amounts of pleural effusion, pericardial effusion, and peritoneal effusion that cannot be controlled by researchers (including but not limited to those that require repeated drainage and have clinical symptoms);
3. Prior to initial administration of anti-tumor therapy: Within 4 weeks or 5 drug half lives (whichever is shorter) prior to administration, anti-tumor drugs (including cytotoxic therapy, targeted therapy, antibody therapy, immunotherapy, etc.) were administered; Received nitrosourea or mitomycin C treatment within 6 weeks prior to administration; Received palliative radiotherapy within 2 weeks prior to administration; Received other anti-tumor treatments such as radical radiotherapy and electric field therapy within 4 weeks before administration; Received traditional Chinese medicine treatment for anti-tumor indications within 2 weeks before administration;
4. Toxic reactions of previous anti-tumor treatments that have not yet improved to CTCAE ≤ 1 (excluding hair loss, skin toxicity, or other toxicity that researchers consider to be of no safety risk);
5. Any situation that affects the ingestion of drugs and seriously affects the absorption or pharmacokinetic parameters of the investigational drug, including but not limited to active gastrointestinal ulcers, long-term gastroesophageal reflux disease (GERD), etc;
6. Severe or uncontrollable heart diseases that require treatment, including any of the following conditions (including but not limited to): ECG QT interval prolongation corrected according to the Fridericia formula, male QTcF>450milliseconds or female QTcF>470milliseconds; Various clinically significant arrhythmias, including but not limited to second degree type II conduction block, third degree conduction block, etc; Cardiac ultrasound indicates a left ventricular ejection fraction (LVEF) of less than 50%; Within 6 months before the first medication, there is myocardial infarction, unstable angina, NYHA class III or IV heart failure; An arterial/venous thrombosis event occurred within 6 months prior to the first medication, and the risk was deemed uncontrollable, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; Or known familial and/or acquired thrombophilia tendencies, such as genetic or acquired defects in anticoagulant proteins, coagulation factors, fibrinolytic proteins, etc; 8 Severe or uncontrolled diabetes (fasting blood glucose ≥ 10mmol/L under the standardized blood pressure reduction program), hypertension (poorly controlled under the standardized blood pressure reduction program, systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg), epilepsy, chronic obstructive pulmonary disease, interstitial pneumonia, pulmonary fibrosis, Parkinson's disease, active bleeding, systemic active infection;

9. Any unstable systemic disease (such as severe liver, kidney, or metabolic diseases such as cirrhosis, renal failure, and uremia); Within 14 days or 5 half lives prior to the first administration, have used CYP3A4 potent and moderate inhibitors and inducers, CYP3A4, CYP2C9, and CYP2C8 sensitive substrates, OATP1B1, OATP1B3, OAT1, OAT3, P-gp, and BCRP substrates (see Appendix 8 for details); 11. Cognitive impairment, history of mental illness, other uncontrolled comorbidities, alcohol dependence, hormone dependence, or drug abuse; Received autologous or allogeneic organ or stem cell transplantation surgery within 3 months prior to the first use of medication; Having undergone major surgery or severe trauma within 4 weeks prior to the first use of medication (excluding biopsy due to sample collection); 13. History of immunodeficiency, including HIV antibody positivity or other acquired or congenital immunodeficiency diseases; 14. There are serious eye diseases (excluding cataracts, etc.), and they have not yet recovered and improved to ≤ level 1; The following serological status reflecting active hepatitis B or hepatitis C infection exists: hepatitis B surface antigen positive or hepatitis B core antibody positive, and HBV DNA>1000 copies/mL; hepatitis C virus antibody positive, and HCV RNA>the upper limit of normal value; 16 cases of active syphilis infection; 17 is known to be severely allergic to the active ingredients or any excipients of the investigational drug; Participated in other clinical trials within 4 weeks prior to the first administration of medication; 19. Patients with positive pregnancy test results or breastfeeding during the screening period; 20 researchers believe that it is not suitable to participate in this study. According to the researchers' assessment, the patient may have other factors that could affect the research results or lead to the forced termination of this study, such as alcohol abuse, drug abuse, other serious illnesses (including mental illnesses) that require concurrent treatment, serious laboratory test abnormalities, and family or social factors that could affect the patient's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2027-08-31 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months.
  Objective Response Rate (ORR) assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST v1.1).

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | From treatment administration up to a maximum duration of 24 months.
  The time from the beginning of the patient's treatment to the disease progression or death for any reason. Based on RECIST criteria v1.1.
Duration of Response(DOR) | Time Frame: Through study completion, an expected average of 24 months
  Duration of Response, from the first time the evaluation results meet CR or PR criteria to the observation of PD or death.
Disease Control Rate (DCR) | From treatment administration up to a maximum duration of 18 months
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD) in total subjects after the last subject participating in.
Overall Survival(OS) | From treatment administration up to a maximum duration of 24 months.
  Overall Survival(OS)
Percentage of Participants With Adverse Events (AEs) | Up to approximately 24 months.
  Number of participants with adverse effects of treatment. Frequency and severity of adverse effects of treatment as assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Ph.D, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
After the completion of the research and academic publication